CLINICAL TRIAL: NCT02798601
Title: Early Induced Hypernatremia for the Prevention and Management of Brain Edema in Patients With Severe Traumatic Brain Injury in a University Hospital
Brief Title: Early Induced Hypernatremia for the Prevention and Management of Brain Edema
Acronym: EHIBE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funds
Sponsor: Hospital Pablo Tobón Uribe (Other)
Collaborators: CES University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U1111-1183-0891; HPTU (Registry Identifier: 2016.049)
Record Dates: First submitted 2016-05-21; First posted 2016-06-14 (Estimated); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Head Trauma
Keywords: Cerebral edema; Hypernatremia; Extended Glasgow Outcome Scale; Intracranial pressure; Mannitol; Hypertonic saline; Mortality
MeSH Terms: conditions — Craniocerebral Trauma; Brain Edema; Hypernatremia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypernatremia (Experimental): Serum sodium between 150 - 155 milliequivalent/L. 7,5% sodium chloride (2 ml/kg every 4 hours), with controls of serum sodium every 4 hours, to achieve a goal of serum sodium between 150 - 155 milliequivalent/L. If after 4 doses of 7.5% sodium chloride the serum sodium is below the target, a bolus of 1 ml/kg of 12% sodium chloride will be used every 4 hours. The goal of serum sodium will be maintained for 48 hours.
  Interventions: Other: Hypernatremia
- Normonatremia (No Intervention): Serum sodium between 135 - 145 milliequivalent/L. Mannitol 100 ml every 4 hours for the first three days; 80 ml every 4 hours the fourth day; 60 ml every 4 hours the fifth day and 40 ml every 4 hours the sixth day and then stopping. The mannitol protocol will be interrupted at any moment if serum sodium is below 135, the systolic blood pressure is below 90 mmHg or the patient has signs of hypovolemia. In this case, 2 ml/kg of 3% sodium chloride every 4 hours will be used until the target of serum sodium is achieved and both, normovolemic state and blood pressure are restored. In addition, the mannitol protocol will be suspended when serum osmolality is above 320.

INTERVENTIONS:
Other: Hypernatremia — Serum Sodium goal: 150 - 155 milliequivalent/L.
  Arms: Hypernatremia

SUMMARY:
The purpose of this study is to estimate the effect of an early induced hypernatremia protocol (150-155 milliequivalent/L) versus normonatremia plus mannitol (135 - 145 milliequivalent/L) in terms of neurologic outcome in patients with severe traumatic brain injury managed at critical care unit.

DETAILED DESCRIPTION:
Severe traumatic brain injury is one of the main causes of death in young people. Additionally, it is considered a public health problem because of the high prevalence of motor and cognitive dysfunction in those who survive.

One of the cornerstones of management is the control of both intracranial pressure and brain edema. It is indicated to use osmotic active solutions to modulate the transit of fluids from the interstitial to the intracellular space. Not only mannitol but also hypertonic saline acts at this point. Currently there is no evidence in favor or against one of them.

Mannitol has been usually recommended for intracranial pressure control in patients with brain trauma. However, others recommend hypertonic saline to achieve a serum sodium level of 160 milliequivalent/L to modulate brain edema. It is not clear if these therapies have an impact on the neurologic prognosis and how frequently adverse effects occur.

ELIGIBILITY:
Inclusion Criteria:

1. Patient greater than 14 years old, who suffered severe non-penetrating Brain Trauma (Glasgow Coma Scale (GCS) equal or less than 8) and a motor GCS equal or less than 5.
2. Criteria time: admitted to the Hospital in the first 24 hours of the Brain Trauma (BT) and admitted to ICU in the first 48 hours of brain trauma.
3. Tomographic evidence of brain edema (one of the following criteria: deviation from the midline, obliteration of perimesencephalic cistern or altered cortico-subcortical differentiation).

Exclusion Criteria:

1. Patient with GCS 3 and bilateral mydriatic pupils and unreactive to light, in the presence of hemodynamic stability (systolic blood pressure equal or greater than 90 mmHg).
2. Patient with insipid diabetes at the ICU admission.
3. Patient with limitation of therapeutic effort.
4. Non-neurological Abbreviated Injury Score greater than 3.
5. Patient past medical history of kidney failure, liver disease or heart failure.
6. Serum sodium less than 135 or greater than 150 milliequivalent/L.
7. Pregnancy.
8. Terminal disease.
9. No authorization to be enrolled in the trial by the patient's caregiver

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01-18 (Estimated); Primary Completion 2017-01-18 (Estimated); Study Completion 2018-01-18 (Estimated)

PRIMARY OUTCOMES:
Glasgow Outcome Scale Extended | 6 months
  The Extended Glasgow Outcome Scale (GOSE) is a global scale for functional outcome that rates patients into eight categories. The categories of severe disability, moderate disability and good recovery are subdivided into a lower and upper category. The scale will be used to evaluate the patient through a phone interview at 6 months of the trauma occurred. The structured interview contains nineteen specific questions which determine upper or lower levels of disability.

SECONDARY OUTCOMES:
All-cause mortality | 28 - day AND 180 - day mortality
  Mortality by any cause
Ventilator - Free Days | 30 days
  Days free of mechanical ventilation at 30 days
Fluid balance. | 5 days
  Net fluid balance (input minus output) (ml) at day 1,2,3,4 y 5.
Acute kidney injury | 7 days
  Acute kidney injury (KDIGO criteria). The criteria for acute kidney injury(AKI) are based on changes in serum creatinine (SCr) and urine output.
  Stage I : Increase in SCr more than 1.5 times baseline, which is known or presumed to have occurred within the prior 7 days OR increase in SCr more than 0.3 mg/dL within 48 hours OR urine output <0.5 ml/kg/h for 6-12h.
  Stage II : Increase in SCr between 2.0 - 2.9 times baseline, which is known or presumed to have occurred within the prior 7 days OR urine output <0.5 ml/kg/h for more than 12 hours.
  Stage III : Increase more than 3.0 times baseline, which is known or presumed to have occurred within the prior 7 days OR Increase in serum creatinine to 4.0 mg/dL OR Initiation of renal-replacement therapy OR urine output <0.3 ml/kg/h for more than 24 hours OR Anuria for more than 12 hours.
Intracranial pressure (ICP) measurement | 5 days
  Intracranial pressure measurement (mmHg) during the first 5 days at the ICU. Estimate the effect of therapies to control intracranial pressure. An intraparenchymal catheter will used to measure the ICP. Intracranial pressure (ICP) will be measured every hour. Intracranial hypertension will be defined as ICP > 20 mm Hg lasting longer than 5 minutes.
Need of second line therapies for brain edema | 7 days
  Secondary decompressive craniectomy or barbituric coma for control of brain edema.
All-cause mortality according to subgroups of monitoring: guided by neurologic examination and serial CT imaging or guided by intracranial pressure monitoring. | 28 - day AND 180 - day mortality
  Estimate the effects of therapies on mortality according to subgroups of treatment (guided by neurologic examination and serial CT imaging or guided by intracranial pressure monitoring).
Glasgow Outcome Scale Extended (GOSE) according to subgroups of monitoring: guided by neurologic examination and serial CT imaging or guided by intracranial pressure monitoring. | 6 Months
  Estimate the effects of therapies on the GOSE according to subgroups of treatment (guided by neurologic examination and serial CT imaging or guided by intracranial pressure monitoring).

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Lopez de Mesa, MD, Principal Investigator — Hospital Pablo Tobon Uribe

IPD SHARING:
Plan to Share IPD: No